CLINICAL TRIAL: NCT01427751
Title: Safety and Efficacy Study of Ozurdex® Compared to Lucentis® in Patients With Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAF-AGN-OPH-RET-004; 2010-023900-29 (EudraCT Number)
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Retinal Vein Occlusion; Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Dexamethasone; Calcium Dobesilate; Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ozurdex® (Active Comparator): Injection of Ozurdex® (dexamethasone intravitreal implant) into the study eye on Day 1 and Month 5. Patients may receive up to one additional treatment, thereafter.
  Interventions: Drug: dexamethasone intravitreal implant
- Lucentis® (Active Comparator): Injection of Lucentis® (ranibizumab) into the study eye on Day 1 and monthly for five months. Patients will receive additional treatment thereafter based on re-treatment criteria.
  Interventions: Biological: ranibizumab

INTERVENTIONS:
Drug: dexamethasone intravitreal implant — Injection of Ozurdex® (dexamethasone intravitreal implant) into the study eye on Day 1 and Month 5. Patients may receive up to one additional treatment, thereafter.
  Other Names: Ozurdex®
  Arms: Ozurdex®
Biological: ranibizumab — Injection of Lucentis® (ranibizumab) into the study eye on Day 1 and monthly for five months. Patients will receive additional treatment thereafter based on re-treatment criteria.
  Other Names: Lucentis®
  Arms: Lucentis®

SUMMARY:
This study will evaluate the safety and efficacy of dexamethasone intravitreal implant (Ozurdex®) compared to ranibizumab (Lucentis®) in patients with branch retinal vein occlusion (BRVO).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of branch retinal vein occlusion in at least one eye
* Visual acuity between 20/400 to 20/40

Exclusion Criteria:

* Active eye infection
* Ocular hypertension which is not controlled on monotherapy (one medication)
* Anticipated need for eye surgery during the study
* Cataract surgery in either eye within 3 months
* Eye surgery including laser of any type within 6 months
* Anti-VEGF treatment in either eye (eg, Lucentis®) within 3 months or systemic anti-VEGF treatment (eg, Avastin) within 6 months
* Use of ocular steroids within 3 months
* Use of steroids (except for inhaled or intranasal) within 1 month or anticipated use during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2014-11-04 (Actual); Study Completion 2014-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (6):
- Paris, France
- Munich, Germany
- Tel Aviv, Israel
- Milan, Italy
- Madrid, Spain
- London, United Kingdom

REFERENCES:
- [Background] Bandello F, Augustin A, Tufail A, Leaback R. A 12-month, multicenter, parallel group comparison of dexamethasone intravitreal implant versus ranibizumab in branch retinal vein occlusion. Eur J Ophthalmol. 2018 Nov;28(6):697-705. doi: 10.1177/1120672117750058. Epub 2018 Apr 9. PMID 29631435

RESULTS

PARTICIPANT FLOW:
Groups:
- Ozurdex®: Injection of Ozurdex® (dexamethasone intravitreal implant) into the study eye on Day 1 and Month 5. Participants may receive up to one additional treatment, thereafter.
- Lucentis®: Injection of Lucentis® (ranibizumab) into the study eye on Day 1 and monthly for five months. Participants will receive additional treatment thereafter based on re-treatment criteria.
Period: Overall Study
Arm/Group | Ozurdex® | Lucentis®
Started | 154 | 153
Completed | 112 | 139
Not Completed | 42 | 14
Not completed — Adverse Event | 18 | 2
Not completed — No further treatment benefit expected | 5 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal of consent | 2 | 2
Not completed — Protocol Violation | 6 | 4
Not completed — Death | 2 | 0
Not completed — Other miscellaneous reasons | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ozurdex® | Lucentis® | Total
Number analyzed (Participants) | 154 | 153 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (10.58) | 65.5 (12.04) | 67.0 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 66 | 128
  Male | 92 | 87 | 179

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: BCVA was measured in the study eye using an eye chart and was recorded as the number of letters read correctly for a total possible score of 0 to 100. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity) A positive change from Baseline (more letters read correctly) indicates improvement.
Time Frame: Baseline, Month 12
Population: Participants from the intent-to-treat population, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ozurdex® | Lucentis®
Number analyzed (Participants) | 154 | 153
letters
  Baseline (n=153,153) | 56.6 (10.89) | 59.2 (10.92)
  Change from Baseline at Month 12 (n=153,151) | 7.9 (14.42) | 16.9 (12.08)

2. Secondary Outcome: Change From Baseline in Central Retinal Subfield Thickness Using Optical Coherence Tomography (OCT)
Description: Optical Coherence Tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina, was performed in the study eye after pupil dilation at Baseline and Month 12. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Month 12
Population: Participants from the intent-to-treat population, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Ozurdex® | Lucentis®
Number analyzed (Participants) | 154 | 153
microns
  Baseline (n=149, 149) | 553.2 (170.15) | 561.0 (188.93)
  Change from Baseline at Month 12 (n=140,144) | -219.2 (180.51) | -253.5 (197.08)

3. Secondary Outcome: Percentage of Patients With 15-or-More Letter Improvement in BCVA
Description: BCVA was measured in the study eye using an eye chart and was recorded as the number of letters read correctly for a total possible score of 0 to 100. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). An improvement in the number of letters read means that the vision has improved.
Time Frame: Baseline, Month 12
Population: Participants from the intent-to-treat population, all randomized participants, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ozurdex® | Lucentis®
Number analyzed (Participants) | 154 | 153
percentage of participants | 33.8 | 59.5

4. Secondary Outcome: Percentage of Patients With a 15-or-More Letter Decrease in BCVA
Description: BCVA was measured in the study eye using an eye chart and was recorded as the number of letters read correctly for a total possible score of 0 to 100. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity).
Time Frame: Baseline, Month 12
Population: Participants from the intent-to-treat population, all randomized participants, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ozurdex® | Lucentis®
Number analyzed (Participants) | 154 | 153
percentage of participants | 9.1 | 0.7

5. Secondary Outcome: Time to BCVA Improvement of 15-or-More Letters
Description: BCVA was measured in the study eye using an eye chart and was recorded as the number of letters read correctly for a total possible score of 0 to 100. The time in days to BCVA improvement of 15-or-More letters.
Time Frame: 12 Months
Population: Participants from the intent-to-treat population, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ozurdex® | Lucentis®
Number analyzed (Participants) | 154 | 153
days | 73.7 (79.68) | 82.0 (93.78)

6. Secondary Outcome: Change From Baseline in National Eye Institute Visual Functioning Questionnaire-25 (VFQ-25)
Description: The VFQ-25 includes 25 vision-targeted questions plus one general health question which assess visual impairment on functioning and specific aspects of health-related quality of life for a total possible composite score of 0 (worst) to 100 (best functionality). A positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 12
Population: Participants from the intent-to-treat population, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozurdex® | Lucentis®
Number analyzed (Participants) | 154 | 153
score on a scale
  Baseline (n=143,139) | 78.1 (16.58) | 80.7 (14.34)
  Change from Baseline at Month 12 (n=143, 139) | 3.5 (12.21) | 6.6 (13.45)

7. Secondary Outcome: Percentage of Participants Not Completing the Month 12 Visit Due to Treatment Failure
Description: Treatment failure was defined as withdrawal of the participant from treatment or from the study by the investigator before the final visit because of a lack of efficacy.
Time Frame: 12 Months
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ozurdex® | Lucentis®
Number analyzed (Participants) | 154 | 153
percentage of participants | 4.5 | 0.7

ADVERSE EVENTS:
Time Frame: Up to 60 Weeks
Description: Safety population, all randomized participants who received at least 1 dose of study drug, was used to determine the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | Ozurdex® | Lucentis®
Serious Adverse Events (participants affected / at risk) | 12/153 | 16/150
Other Adverse Events (participants affected / at risk) | 127/153 | 104/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ozurdex® (N=153) | Lucentis® (N=150)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Agitated depression (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Catheter site related reaction (General disorders) | 0 | 1
Ocular hypertension (Eye disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Endophthalmitis (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ozurdex® (N=153) | Lucentis® (N=150)
Conjunctival haemorrhage (Eye disorders) | 28 | 17
Macular oedema (Eye disorders) | 20 | 4
Visual acuity reduced (Eye disorders) | 18 | 3
Cataract (Eye disorders) | 13 | 2
Lenticular opacities (Eye disorders) | 10 | 0
Ocular hypertension (Eye disorders) | 9 | 1
Blepharitis (Eye disorders) | 9 | 3
Dry eye (Eye disorders) | 9 | 7
Vitreous floaters (Eye disorders) | 9 | 9
Eye pain (Eye disorders) | 6 | 9
Conjunctivitis (Eye disorders) | 6 | 9
Intraocular pressure increased (Investigations) | 50 | 16
Nasopharyngitis (Infections and infestations) | 8 | 5
Headache (Nervous system disorders) | 4 | 9
Hypertension (Vascular disorders) | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to release and can embargo communications regarding trial results for a period that is less than or equal to 120 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.